CLINICAL TRIAL: NCT01043783
Title: Preliminary Data for Breath Biofeedback of Dietary Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M-2009-1107
Record Dates: First submitted 2009-12-15; First posted 2010-01-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dietary Adherence — Subjects consumed a specified healthy, balanced, reduced calorie diet and provided timed breath samples.

SUMMARY:
The investigators ultimate goal is to test the hypothesis that immediate feedback of dietary adherence will enhance compliance to a weight loss program. This study deals directly with gathering the needed preliminary data for a grant submission.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females age 18 or older

Exclusion Criteria:

* Chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Breath CO2, ketones, aldehydes, alcohols | Daily for 5-7 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States